CLINICAL TRIAL: NCT04734782
Title: Assess the Correlation With Severe Respiratory Syncytial Virus Disease in the First 6 Months in Children With Congenital Heart Disease and Maternal Ac-AntiVSR Titers During Pregnancy
Acronym: (VSRyCC)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Angeles Lomas (Other)
Responsible Party: Principal Investigator, Humberto Garcia Aguilar, Master in Science, Hospital Angeles Lomas
Other Study IDs: 025.2021
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Syncytial Virus, Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protective Mothers (high IGG titers): Protected group Newborns with congenital heart disease + high titers of anti-RSV IGG in the mother's serum before birth
  Interventions: Diagnostic Test: Determination of antibodies in maternal serum IgG for respiratory syncytial virus
- Non-protective mothers (low IGG titers): Unprotected group Newborn with congenital heart disease + negative anti-RSV IGG titers in the mother's serum before birth.
  Interventions: Diagnostic Test: Determination of antibodies in maternal serum IgG for respiratory syncytial virus

INTERVENTIONS:
Diagnostic Test: Determination of antibodies in maternal serum IgG for respiratory syncytial virus — By venipuncture, a blood sample will be taken and the levels of anti-RSV IgG antibodies will be processed in serum by commercial techniques.

SUMMARY:
Passive transplacental immunity against the respiratory syncytial virus (RSV) appears to mediate infant protection during the first 6 months of life (1). Observations of environmental exposure in pregnant women during an RSV epidemic could influence these children's susceptibility to infection by offering levels of antibodies that are transferred to the fetus. However, there is no prospective study in the population at risk such as children with congenital heart disease, as well as the effective levels of anti-RSV immunoglobulin G (IgG) as protective biomarkers for RSV infection after delivery (2)

Justification

The most serious evolution of the clinical disease of acute RSV bronchiolitis in children under 6 months of age is related to lower exposure of the pregnant woman to the RSV epidemic. With maternal immunization through natural exposure, it is logical to relate protection to children for severe RSV disease. However, it is not proven (3).

1. - Nandapalan N, Taylor CE, Greenwell J, et al. Seasonal variations in maternal serum and mammary immunity to RS virus. J Med Virol. 1986;20(1):79-87. doi:10.1002/jmv.1890200110
2. - Stensballe LG, Ravn H, Kristensen K, Meakins T, Aaby P, Simoes EA. Seasonal variation of maternally derived respiratory syncytial virus antibodies and association with infant hospitalizations for respiratory syncytial virus. J Pediatr. 2009;154(2):296-298. doi:10.1016/j.jpeds.2008.07.053
3. - Ramos-Fernández JM, et al. Does exposure of pregnant women to epidemic respiratory syncytial virus affect the severity of bronchiolitis? Enferm Infec Microbiol Clin. 2017. https://doi.org/10.1016/j.eimc.2018.07.002)

DETAILED DESCRIPTION:
A prospective cohort study of mothers with a prenatal diagnosis of a fetus with congenital heart disease will be carried out. To whom titers will be measured. Anti-RSV IGG antibodies result from previous exposure.

According to the IGG titers in anti-RSV serum, 2 groups will be formed:

Protective Mothers (high IGG titers) Non-protective mothers (low IGG titers) The products will be followed up for 6 months after birth to correlate the maternal titers of Ac anti-RSV with the presence and severity of respiratory infection by RSV (Bronchiolitis) in this period.

Population and period

Pregnant women evaluated in the National Medical Center 20 de Noviembre, Pediatric Cardiology service for the prenatal diagnosis of congenital heart disease in their fetuses. Newborns with corroborated congenital heart disease with prenatal diagnosis.

Study inclusion period February 1, 2021, to October 30, 2021. Study follow-up period March 1 2021 to December 30 2021.

Sample type: Non-randomized, for convenience, sequential and with an estimated of 30 patients per group.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant mothers in the third trimester of gestational age, with a child with congenital heart disease diagnosed by fetal echocardiogram
2. Approval of informed consent
3. Newborn of term or preterm, with corroborated congenital heart disease and presenting with a respiratory infection by RSV

Exclusion Criteria:

1. - Non-acceptance of informed consent
2. - Premature birth and need for neonatal intensive care for more than 4 weeks.
3. - Newborn with bronchopulmonary dysplasia

Elimination criteria

1.- Use of palivizumab

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pregnant women evaluated in the National Medical Center 20 de Noviembre, Pediatric Cardiology service for the prenatal diagnosis of congenital heart disease in their fetuses. Newborns with corroborated congenital heart disease with prenatal diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Determination of antibodies in maternal serum IgG for respiratory syncytial virus | 12 months
  By venipuncture, a blood sample will be taken and the levels of anti-RSV IgG antibodies will be processed in serum by commercial techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Nacional 20 de Noviembre, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon direct request with the principal investigator through official and unofficial communication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years